CLINICAL TRIAL: NCT04798196
Title: Using Smart Devices to Implement an Evidence-based eHealth System for Older Adults
Brief Title: ElderTree Smart System for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020-0868; A195000 (Other: UW Madison); Protocol Version 10/20/2021 (Other: UW Madison); ENGR/INDUSTRIAL ENGR (Other: UW Madison); 1R18HS026853-01A1 (AHRQ)
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Chronic Pain
Keywords: Chronic conditions; Voice-activated "smart" technology
MeSH Terms: conditions — Chronic Pain; Chronic Disease | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): Participants will receive treatment as usual (TAU).
  Interventions: Behavioral: Treatment as usual (TAU)
- ElderTree on laptop (ET- LT) (Experimental): Participants will receive ElderTree on a laptop.
  Interventions: Behavioral: ElderTree on laptop (ET- LT)
- ElderTree on smart system (ET- SS) (Experimental): Participants will receive ElderTree on a smart system.
  Interventions: Behavioral: ElderTree on smart system (ET- SS)

INTERVENTIONS:
Behavioral: ElderTree on laptop (ET- LT) — ElderTree (ET) is an existing intervention providing tools, motivation, and support on a computer platform to help older adults manage their health.
  ET is based on the extensively tested Comprehensive Health Enhancement Support System (CHESS). ET is a "walled garden" free of ads, with design features based on older users' feedback as well as best-practice principles such as uncluttered screens and large type. ET uses computers to deliver key elements of successful interventions: long duration, ongoing outreach, prompts, monitoring, cognitive reframing, action planning, problem solving, self-tailoring, and peer support. ET-LT arm will access ET on Laptop (ET- LT)
  Arms: ElderTree on laptop (ET- LT)
Behavioral: ElderTree on smart system (ET- SS) — ElderTree (ET) is an existing intervention providing tools, motivation, and support on a computer platform to help older adults manage their health.
  ET is based on the extensively tested Comprehensive Health Enhancement Support System (CHESS). ET is a "walled garden" free of ads, with design features based on older users' feedback as well as best-practice principles such as uncluttered screens and large type. ET uses computers to deliver key elements of successful interventions: long duration, ongoing outreach, prompts, monitoring, cognitive reframing, action planning, problem solving, self-tailoring, and peer support.
  ElderTree on smart system (ET- SS) will use voice-activated "smart" speakers connected to the Internet. Because they are used by talking and listening rather than typing and reading, many barriers associated with laptop use can be avoided.
  Arms: ElderTree on smart system (ET- SS)
Behavioral: Treatment as usual (TAU) — Treatment as usual (TAU)
  Arms: Control group

SUMMARY:
Multiple chronic conditions (MCCs) are costly and pervasive among older adults. MCCs account for 90% of Medicare spending, and 65% of Medicare beneficiaries have 3 or more chronic conditions; 23% have 5 or more. MCCs are often addressed in primary care, where time pressures force a focus on medication and lab results rather than self-management skills.

The primary purpose of this study is to investigate whether voice-activated "smart" technology increases adoption and sustains use of an evidence-based electronic health intervention (Elder Tree, or ET) for older adults with multiple chronic conditions, and thereby improves its potential to widely enhance quality of life and health outcomes. ET is an existing intervention providing tools, motivation, and support on a computer platform to help older adults manage their health.

An Agency for Health Care Research and Quality (AHRQ)-funded randomized controlled trial (RCT) found that ET improved quality of life and other factors among high users of primary care with multiple chronic conditions such as diabetes and hypertension. However, many people did not use it extensively, which is a common problem with all web apps.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥60 years old;
* Have been treated in University of Wisconsin (UW) Health clinics, with no plans to leave during the study period (only relevant for UW Health patients, not patients recruited from the community);
* Have a chronic pain diagnosis AND a medical diagnoses of three or more of the following common chronic conditions: Chronic obstructive pulmonary disease (COPD), asthma, diabetes, hyperlipidemia, hypertension, ischemic heart disease, atrial fibrillation, heart failure, stroke, BMI 30+, cancer, chronic kidney disease, depression, osteoporosis, arthritis, or dizziness/falls/loss of vestibular function;
* Be willing to share healthcare use (e.g. 30-day readmissions) in electronic health records (only relevant for UW Health patients, not patients recruited from the community); and
* Allow researchers to share information about a patient's health status with their primary care physician (PCP).

Exclusion Criteria:

* Require an interpreter
* Have a medical diagnosis of any of the following:

  * Alzheimer's
  * Schizophrenia/other psychotic disorders
  * Dementia
  * Autism spectrum disorder
  * Known terminal illness with less than 6 months to live
  * Acute medical problem requiring immediate hospitalization

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Gustafson, PhD, Principal Investigator — UW-Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Landucci G, Gustafson DH Sr, Mares ML, Pe-Romashko K, Curtin JJ, Hu Y, Maus A, Thompson K, Saunders S, Brown K, Woodburn J, Mutlu B. Using Smart Displays to Implement an eHealth System for Older Adults With Multiple Chronic Conditions: Randomized Controlled Trial. JMIR Aging. 2025 Nov 18;8:e75991. doi: 10.2196/75991. PMID 40961249
- [Derived] Gustafson DH Sr, Mares ML, Johnston DC, Landucci G, Pe-Romashko K, Vjorn OJ, Hu Y, Gustafson DH Jr, Maus A, Mahoney JE, Mutlu B. Using Smart Displays to Implement an eHealth System for Older Adults With Multiple Chronic Conditions: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 May 5;11(5):e37522. doi: 10.2196/37522. PMID 35511229

RESULTS

PARTICIPANT FLOW:
Groups:
- ElderTree on Laptop (ET- LT): Participants will receive ElderTree on a laptop.
  ElderTree on laptop (ET- LT): ElderTree (ET) is an existing intervention providing tools, motivation, and support on a computer platform to help older adults manage their health.
  ET is based on the extensively tested Comprehensive Health Enhancement Support System (CHESS). ET is a "walled garden" free of ads, with design features based on older users' feedback as well as best-practice principles such as uncluttered screens and large type. ET uses computers to deliver key elements of successful interventions: long duration, ongoing outreach, prompts, monitoring, cognitive reframing, action planning, problem solving, self-tailoring, and peer support. ET-LT arm will access ET on Laptop (ET- LT)
- ElderTree on Smart System (ET- SS): Participants will receive ElderTree on a smart system.
  ElderTree on smart system (ET- SS): ElderTree (ET) is an existing intervention providing tools, motivation, and support on a computer platform to help older adults manage their health.
  ET is based on the extensively tested Comprehensive Health Enhancement Support System (CHESS). ET is a "walled garden" free of ads, with design features based on older users' feedback as well as best-practice principles such as uncluttered screens and large type. ET uses computers to deliver key elements of successful interventions: long duration, ongoing outreach, prompts, monitoring, cognitive reframing, action planning, problem solving, self-tailoring, and peer support.
  ElderTree on smart system (ET- SS) will use voice-activated "smart" speakers connected to the Internet. Because they are used by talking and listening rather than typing and reading, many barriers associated with laptop use can be avoided.
Period: Overall Study
Arm/Group | Control Group | ElderTree on Laptop (ET- LT) | ElderTree on Smart System (ET- SS)
Started | 91 | 91 | 86
4 Month Time Point | 86 | 86 | 77
8 Month Time Point | 84 | 85 | 80
Completed | 88 | 90 | 83
Not Completed | 3 | 1 | 3
Not completed — Lost to Follow-up | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- ElderTree on Laptop (ET- LT): Participants will receive ElderTree on a laptop.
  ElderTree on laptop (ET- LT): ElderTree (ET) is an existing intervention providing tools, motivation, and support on a computer platform to help older adults manage their health.
- ElderTree on Smart System (ET- SS): Participants will receive ElderTree on a smart system.
  ElderTree (ET) is an existing intervention providing tools, motivation, and support on a computer platform to help older adults manage their health.
  ElderTree on smart system (ET- SS) will use voice-activated "smart" speakers connected to the Internet. Because they are used by talking and listening rather than typing and reading, many barriers associated with laptop use can be avoided.
- Total: Total of all reporting groups
Arm/Group | Control Group | ElderTree on Laptop (ET- LT) | ElderTree on Smart System (ET- SS) | Total
Number analyzed (Participants) | 91 | 91 | 86 | 268
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.49 (7.77) | 69.76 (7.39) | 70.13 (6.86) | 69.79 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 59 | 55 | 177
  Male | 28 | 32 | 31 | 91
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Participants: Asian | 0 | 1 | 0 | 1
  Participants: Black or African American & American Indian or Alaskan Native | 2 | 1 | 0 | 3
  Participants: Black, Euro-African, or African American | 20 | 16 | 14 | 50
  Participants: White | 68 | 72 | 71 | 211
  Participants: White & Hispanic or Latino | 1 | 1 | 0 | 2
  Participants: White, Black or African American, & American Indian or Alaskan Native | 0 | 0 | 1 | 1
Number of chronic conditions [Mean (Standard Deviation); unit: chronic conditions] — Number of chronic conditions was reported by participants from a list of 17 chronic conditions: chronic pain, COPD, asthma, diabetes, high cholesterol, high blood pressure, ischemic heart disease (coronary heart or coronary artery disease), atrial fibrillation, heart failure, stroke, BMI 30+, cancer, chronic kidney disease, depression, osteoporosis, arthritis, and dizziness/falls/loss of vestibular function.
  chronic conditions | 6.52 (2.31) | 6.54 (2.54) | 6.57 (2.55) | 6.54 (2.46)

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v2.1 - Pain Interference Score
Description: Pain interference was measured using the 4-item subscale from the PROMIS 29. The items asked participants to answer regarding the past 7 days. Scoring of individual items varies and is calculated by the scale's developers; with higher values indicating more pain interference. The possible range is 41.1 to 76.3 (PROMIS scores reported here have weighted ranges).
Time Frame: Baseline, 4 months, 8 months
Population: All participants did not return surveys at 4 and 8 month time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- ElderTree on Smart System (ET- SS): Participants will receive ElderTree on a smart system.
  ElderTree on smart system (ET- SS): ElderTree (ET) is an existing intervention providing tools, motivation, and support on a computer platform to help older adults manage their health.
  ElderTree on smart system (ET- SS) will use voice-activated "smart" speakers connected to the Internet. Because they are used by talking and listening rather than typing and reading, many barriers associated with laptop use can be avoided.
Arm/Group | Control Group | ElderTree on Laptop (ET- LT) | ElderTree on Smart System (ET- SS)
Number analyzed (Participants) | 91 | 91 | 86
score on a scale
  Baseline | 58.44 (7.98) | 59.57 (7.83) | 59.19 (7.86)
  4 months: number analyzed (Participants) | 86 | 86 | 77
  4 months | 57.94 (8.88) | 58.20 (7.55) | 57.99 (7.39)
  8 months: number analyzed (Participants) | 84 | 85 | 80
  8 months | 57.50 (9.39) | 57.63 (7.88) | 57.77 (8.31)

2. Primary Outcome: Change in PROMIS Short Form v2.1 - Psychosocial Quality of Life Score
Description: Psychosocial quality of life was measured using the 12-item subscale from the PROMIS 29. The items asked participants to answer regarding the past 7 days. Scoring of individual items varies and is calculated by the scale's developers; with higher values indicating better quality of life. The possible range is 21.2 to 67.6.
Time Frame: Baseline, 4 months, 8 months
Population: All participants did not return surveys at 4 and 8 month time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | ElderTree on Laptop (ET- LT) | ElderTree on Smart System (ET- SS)
Number analyzed (Participants) | 91 | 91 | 86
score on a scale
  Baseline | 46.40 (7.26) | 45.26 (7.95) | 46.50 (7.81)
  4 months: number analyzed (Participants) | 86 | 86 | 77
  4 months | 46.11 (8.34) | 46.29 (7.98) | 46.88 (7.12)
  8 months: number analyzed (Participants) | 84 | 85 | 80
  8 months | 47.20 (7.88) | 45.81 (8.26) | 47.02 (7.72)

3. Secondary Outcome: ElderTree Days of Use
Description: Days of ElderTree use within a 4 month period before their survey date. The possible range for days of ElderTree use is 0 to 120.
Time Frame: baseline to 4 months, and 4 months to 8 months
Population: The control group did not use ElderTree, all participants did not return surveys at 4 and 8 month time points.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Control Group | ElderTree on Laptop (ET- LT) | ElderTree on Smart System (ET- SS)
Number analyzed (Participants) | 0 | 91 | 86
Days
  Baseline to 4 months: number analyzed (Participants) | 0 | 86 | 77
  Baseline to 4 months |  | 28.47 (19.28) | 19.02 (16.09)
  4 months to 8 months: number analyzed (Participants) | 0 | 86 | 77
  4 months to 8 months |  | 17.48 (14.34) | 10.08 (9.85)

4. Secondary Outcome: Physical Quality of Life
Description: Physical quality of life was measured using the 12-item subscale from the PROMIS 29 (Patient-Reported Outcomes Measurement Information System) Global Health. The items asked participants to answer regarding the past 7 days. Scoring of individual items varies and is calculated by the scale's developers; with higher values indicating more physical quality of life. The possible range is 16.2-67.7.
Time Frame: Baseline, 4 months, 8 months
Population: All participants did not return surveys at 4 and 8 month time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | ElderTree on Laptop (ET- LT) | ElderTree on Smart System (ET- SS)
Number analyzed (Participants) | 91 | 91 | 86
score on a scale
  Baseline | 40.23 (9.23) | 40.84 (9.11) | 41.01 (8.35)
  4 months: number analyzed (Participants) | 86 | 86 | 77
  4 months | 40.28 (9.61) | 41.30 (9.15) | 41.65 (8.30)
  8 months: number analyzed (Participants) | 84 | 85 | 80
  8 months | 40.36 (10.04) | 40.89 (9.55) | 42.12 (8.67)

5. Secondary Outcome: Pain Intensity
Description: Pain intensity was measured using a single item subscale from the PROMIS 29 (Patient-Reported Outcomes Measurement Information System) Global Health. The item asked participants to answer regarding the past 7 days. The raw score of the item was used (range: 0-10); with higher values indicating more pain intensity.
Time Frame: Baseline, 4 months, 8 months
Population: All participants did not return surveys at 4 and 8 month time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | ElderTree on Laptop (ET- LT) | ElderTree on Smart System (ET- SS)
Number analyzed (Participants) | 91 | 91 | 86
units on a scale
  Baseline | 4.48 (2.27) | 4.53 (2.07) | 4.64 (2.27)
  4 Months: number analyzed (Participants) | 86 | 86 | 77
  4 Months | 4.21 (2.29) | 4.13 (1.91) | 4.39 (2.43)
  8 Months: number analyzed (Participants) | 84 | 85 | 80
  8 Months | 4.00 (2.38) | 4.09 (2.11) | 4.58 (2.57)

6. Secondary Outcome: Number of Participants Readmitted Within 30-days
Description: 30-day readmissions were measured using a single item asking participants to answer regarding the past 4 months. The raw score, answering yes/no to having a 30-day readmission, was used. Those participants answering 'yes' to being readmitted in the last 30 days are reported for each time point.
Time Frame: Baseline, 4 months, 8 months
Population: All participants did not return surveys at 4 and 8 month time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | ElderTree on Laptop (ET- LT) | ElderTree on Smart System (ET- SS)
Number analyzed (Participants) | 91 | 91 | 86
Participants
  Baseline | 4 | 4 | 5
  4 months: number analyzed (Participants) | 86 | 86 | 77
  4 months | 5 | 6 | 3
  8 months: number analyzed (Participants) | 84 | 85 | 80
  8 months | 7 | 5 | 6

7. Secondary Outcome: Health Distress
Description: Health distress was measured using the 4-item Lorig Health Distress Scale. The items asked participants to answer regarding the past month. The measure was scored by averaged the items; with higher values indicating more health distress. Possible range is 0 to 5.
Time Frame: Baseline, 4 months, 8 months
Population: All participants did not return surveys at 4 and 8 month time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | ElderTree on Laptop (ET- LT) | ElderTree on Smart System (ET- SS)
Number analyzed (Participants) | 91 | 91 | 86
score on a scale
  Baseline | 2.02 (1.32) | 2.04 (1.20) | 1.88 (1.28)
  4 months: number analyzed (Participants) | 86 | 86 | 77
  4 months | 1.78 (1.32) | 1.85 (1.24) | 1.71 (1.21)
  8 months: number analyzed (Participants) | 84 | 85 | 80
  8 months | 1.68 (1.24) | 1.93 (1.21) | 1.62 (1.10)

8. Secondary Outcome: Well-being
Description: Well-being was measured using the 5-items World Health Organization (WHO) Well-Being Index. The items asked participants to answer regarding the past 7 days. The measure was scored by summing the items; with higher values indicating better well-being. Possible range is 0 to 25.
Time Frame: Baseline, 4 months, 8 months
Population: All participants did not return surveys at 4 and 8 month time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | ElderTree on Laptop (ET- LT) | ElderTree on Smart System (ET- SS)
Number analyzed (Participants) | 91 | 91 | 86
score on a scale
  Baseline | 12.75 (5.55) | 12.56 (5.74) | 13.12 (5.81)
  4 months: number analyzed (Participants) | 86 | 86 | 77
  4 months | 13.20 (5.93) | 13.21 (5.42) | 13.48 (5.31)
  8 months: number analyzed (Participants) | 84 | 85 | 80
  8 months | 13.27 (5.78) | 12.80 (5.69) | 14.15 (5.87)

9. Secondary Outcome: Loneliness
Description: Loneliness was measured using the 5-item NIH Toolbox Social Relationship Scale Loneliness. The items asked participants to answer regarding the past month. Scoring of individual items varies and is calculated by the scale's developers; with higher values indicating more Loneliness. Possible range is 20 to 80.
Time Frame: Baseline, 4 months, 8 months
Population: All participants did not return surveys at 4 and 8 month time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | ElderTree on Laptop (ET- LT) | ElderTree on Smart System (ET- SS)
Number analyzed (Participants) | 91 | 91 | 86
score on a scale
  Baseline | 52.93 (11.76) | 55.19 (12.55) | 53.49 (13.32)
  4 months: number analyzed (Participants) | 86 | 86 | 77
  4 months | 51.41 (12.63) | 55.13 (11.63) | 52.45 (12.86)
  8 months: number analyzed (Participants) | 84 | 85 | 80
  8 months | 51.60 (12.85) | 53.84 (12.12) | 50.51 (12.16)

10. Secondary Outcome: Irritability
Description: Irritability was measured using the 5-item Brief Irritability Test. The items asked participants to answer regarding the past 7 days. The measure was scored by summing the items; with higher values indicating more irritability. Possible range is 5 to 30.
Time Frame: Baseline, 4 months, 8 months
Population: All participants did not return surveys at 4 and 8 month time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | ElderTree on Laptop (ET- LT) | ElderTree on Smart System (ET- SS)
Number analyzed (Participants) | 91 | 91 | 86
score on a scale
  Baseline | 11.30 (4.32) | 11.13 (4.14) | 10.59 (4.66)
  4 months: number analyzed (Participants) | 86 | 86 | 77
  4 months | 10.70 (4.01) | 10.72 (4.05) | 10.22 (4.41)
  8 months: number analyzed (Participants) | 84 | 85 | 80
  8 months | 10.38 (4.25) | 10.45 (4.20) | 9.65 (3.95)

11. Secondary Outcome: Communication With Physicians
Description: Communication with physicians was measured using the 3-item Lorig Communication with Physicians. The items asked participants to answer regarding the past 4 months. The measure was scored by averaging the items; with higher values indicating better communication with the healthcare provider. Possible range is 0 to 5.
Time Frame: Baseline, 4 months, 8 months
Population: All participants did not return surveys at 4 and 8 month time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | ElderTree on Laptop (ET- LT) | ElderTree on Smart System (ET- SS)
Number analyzed (Participants) | 91 | 91 | 86
score on a scale
  Baseline | 3.16 (1.20) | 3.11 (1.08) | 2.93 (1.35)
  4 months: number analyzed (Participants) | 86 | 86 | 77
  4 months | 3.22 (1.39) | 3.37 (1.15) | 3.42 (1.05)
  8 months: number analyzed (Participants) | 84 | 85 | 80
  8 months | 3.26 (1.47) | 3.18 (1.39) | 3.29 (1.20)

ADVERSE EVENTS:
Time Frame: 8 months
Description: Adverse events in Redcap
Arm/Group | Control Group | ElderTree on Laptop (ET- LT) | ElderTree on Smart System (ET- SS)
All-Cause Mortality (participants affected / at risk) | 3/91 | 1/91 | 1/86
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/91 | 0/86
Other Adverse Events (participants affected / at risk) | 0/91 | 0/91 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT04798196/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT04798196/ICF_001.pdf